CLINICAL TRIAL: NCT02548897
Title: Uncovering an Electrical Biomarker for Freezing of Gait in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB201500458
Record Dates: First submitted 2015-09-10; First posted 2015-09-14 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease with Freezing of Gait Symptoms
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Freezing of gait in PD (Experimental): All participants will undergo an deep brain stimulation (DBS) for the FOG, and an electroencephalography (EEG) to better understand the neurophysiological underpinnings of the symptom. In addition, review changes in scalp recorded EEG and gait parameters during natural FoG episodes while participants are ambulatory in an advanced gait laboratory setting using a wireless EEG amplifier with active electrodes.
  Interventions: Device: Deep brain stimulation; Other: Electroencephalography

INTERVENTIONS:
Device: Deep brain stimulation — The programming of DBS settings in all participants with bilateral DBS implants in the globus pallidus internus (GPi) and pedunculopontine nucleus (PPN) will be performed.
  Other Names: DBS
Other: Electroencephalography — An electroencephalography (EEG) will be performed on all participants to better understand the neurophysiological underpinnings of the symptom.
  Other Names: EEG

SUMMARY:
The purpose of this study is to investigate brain signals related to freezing of gait (FoG), a symptom of Parkinson's Disease, that can lead to dangerous falls. The investigators hypothesize that uncovering these signals can lead to better deep brain stimulation interventions.

DETAILED DESCRIPTION:
Freezing of gait (FoG) is a devastating symptom of Parkinson's disease (PD) that affects more than half of the patient population. Defined as an intermittent failure to initiate or maintain effective stepping, FoG is a common cause of falls and injuries in PD. There is an unmet but pressing need to develop novel therapeutic strategies to treat disabling drug- and deep brain stimulation (DBS)-resistant FoG in PD. The objective of this research study is to uncover an electrical biomarker for FoG from human electroencephalography (EEG) to better understand the neurophysiological underpinnings of the symptom and to inform the development of clinical interventions for FoG. The central hypothesis is that EEG activity over the motor cortex will exhibit significant changes leading up to and during FoG episodes. This biomarker can then facilitate the detection of FoG events directly from scalp recordings. The rationale for the proposed research is that non-invasive detection of FoG episodes can be used to guide responsive DBS strategies to resolve the episode and prevent potential injuries. Furthermore, it is hypothesize that this biomarker will modulate when therapeutic DBS settings for FoG are turned on. Given the vast number of DBS parameter combinations that need to be tested and chronically verified, such a biomarker can significantly shorten clinical programming and prevent side effects of non-optimal stimulation settings. This study will review changes in scalp recorded EEG and gait parameters during natural FoG episodes while participants are ambulatory in an advanced gait laboratory setting using a wireless EEG amplifier with active electrodes. The modulation of the uncovered biomarker during clinical programming of DBS settings in participants with bilateral DBS implants in the globus pallidus internus (GPi) and pedunculopontine nucleus (PPN). This project is innovative as the dataset acquired will be the first of its kind in PD patients with FoG, and will open a new direction of multidisciplinary investigation that can potentially uncover the cortical mechanisms of FoG in humans and which in turn could lead to novel and effective therapies for those suffering from PD. This contribution will be significant because it will provide a critical and unmet therapeutic option for FoG and decrease morbidity and mortality associated with FoG related falls.

In summary, the following goals will be accomplished:

* Recruit subjects who have undergone DBS implantation for the treatment of PD and who have clinically verified FoG.
* Collect EEG data during ambulatory tasks that often induce FoG episodes and uncover biomarkers of FoG.
* Develop a closed-loop paradigm for acute testing when FoG events are detected from EEG data.
* Use the EEG biomarkers to guide DBS parameter selection for treatment of FoG.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of idiopathic PD, without a previous DBS operation and must be deemed appropriate for a DBS operation by the interdisciplinary screening team (must meet UK Brain Bank criteria for diagnosis of idiopathic Parkinson's disease).
* Experiencing significant gait and postural instability despite optimal pharmacologic management (Hoehn and Yahr Stage II or greater in the on state).
* Best medication "on" does not reveal meaningful improvement in posture scores (Pull Test). Patients must be challenged in person with a suprathreshold dose of levodopa (1.5 times optimized regular dose of levodopa) and must have poor or no improvement in postural stability.
* Patients must possess a clinical history of gait freezing > 2 episodes per month, to be included, participants must also score > 1 on item #3 of the Freezing of Gait (FOG) Questionnaire and exhibit five or more FoG episodes during the provocation protocol in on or off state.
* L-dopa responsive with clearly defined "on" periods.
* Willingness and ability to cooperate during conscious operative procedure, as well as during post-surgical evaluations, adjustments of medications and stimulator settings.

Exclusion Criteria:

* Clinically significant medical disease that would increase the risk of developing pre- or postoperative complications. Clinically significant medical disease includes uncontrolled systemic hypertension with values above 170/100mmHg; cardiac or pulmonary disease; uncorrected coagulation abnormalities or need for therapeutic anticoagulation which cannot be interrupted; any condition that would render the patient unable to safely cooperate with the study tests as judged by the screening physician.
* Evidence of secondary or atypical parkinsonism.
* Other neurological and musculoskeletal impairments that would negatively influence postural stability
* Past MRI scan with significant evidence of brain atrophy or other abnormalities.
* Dementia as evidenced by impairment in two neuropsychological domains and a Mattis Dementia Score <130.
* A major untreated psychiatric disorder as revealed on psychiatric exam at screening, and a Beck Depression Inventory Score >14.
* Subjects with a history of seizures.
* Subjects who may require repeat MRI scans.
* Subjects with a history of a cranial neurosurgical procedure.
* Subjects with metal in the head or another implanted stimulator (e.g. vagus nerve stimulator, spinal cord stimulator, pacemaker, cochlear implant, etc).
* Subjects who require treatment with Electroconvulsive therapy (ECT) or repetitive Transcranial Magnetic Stimulation (rTMS).
* Pregnant or nursing women or women who wish to become pregnant will be excluded.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-10; Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Number of freezing of gait events | up to months 24 post DBS surgery

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Gunduz, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States